CLINICAL TRIAL: NCT01271023
Title: Inpatient Evaluation of an Automated Closed-Loop Control-to-Range System
Acronym: CTR
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Responsible Party: Principal Investigator, John Lum, Principal Investigator, Jaeb Center for Health Research
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTR
Record Dates: First submitted 2011-01-04; First posted 2011-01-06 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-09

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Closed-Loop Control (Experimental): The Control to Range algorithm will be used in conjunction with continuous glucose monitoring and insulin pump delivery to manage the subject's blood glucose.
  Interventions: Device: Control-to-Range Automated Insulin Management System

INTERVENTIONS:
Device: Control-to-Range Automated Insulin Management System — The devices that will be used in the Closed-Loop Control System are standardized across all study sites and include the DexCom Seven Plus Continuous Glucose Monitor (CGM), the OmniPod insulin pump, and the FreeStyle blood glucose meter. The Closed-Loop Control System will be used during all 3 admission visits.

SUMMARY:
The purpose of this study is to test an insulin management system ("Control-to-Range (CTR) system") in an inpatient setting to see if the system is safe and effective enough to test in a future at-home study. The system includes (1) a DexCom Seven Plus Continuous Glucose Monitoring (CGM) device that measures the blood sugar, (2) a laptop computer that determines how much insulin is needed, and (3) an Insulet OmniPod insulin pump that delivers the insulin.

The study will include two hospital stays consisting of meals and exercise scenarios. Both hospital stays will be for 24+ hours during the day and night. The study will include about 50 individuals at 7 clinical centers in the United States, France, Israel, and Italy.

DETAILED DESCRIPTION:
Clinical Research Center (CRC) Session Detail (closed-loop control active for all elements)

Day 1 (24+ hours):

1. Admission at 7:00 AM
2. Standardized breakfast with normal bolus at 9:00 AM
3. Lunch with normal bolus at 1:00 PM
4. Dinner with normal bolus at 7:00 PM
5. Overnight sleep
6. Breakfast with missed meal bolus followed by user alert and correction bolus
7. Discharge

Day 2 (24+ hours):

1. Admission at 7:00 AM
2. Standardized breakfast with normal bolus at 9:00 AM
3. Lunch with normal bolus at 1:00 PM
4. Exercise
5. Dinner with normal bolus at 7:00 PM
6. Overnight sleep
7. Breakfast with overbolus at 7:00 AM
8. Discharge

Meal boluses will be semi-automated, with manual meal announcement by the physician/nurse, automated bolus recommendation by the system, and automated delivery of the bolus following confirmation of the recommendation. Between-meal insulin dosing will be fully automated; bolus confirmation by the physician/nurse will be requested by the closed-loop controller only when it determines that carbohydrates may be necessary to avoid hypoglycemia following the bolus.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of type 1 diabetes for at least one year and using an insulin pump for at least 6 months The diagnosis of type 1 diabetes is based on the investigator's judgment; C peptide level and antibody determinations are not needed.
* Age 12 to 65 years
* Hemoglobin A1c (HbA1c) between 5.0% and 10.5%, as measured with DCA2000 or equivalent device
* For females, not currently known to be pregnant
* Demonstration of proper mental status and cognition for the study
* An understanding of and willingness to follow the protocol and sign the informed consent or assent

Exclusion Criteria:

* Diabetic ketoacidosis in the past 6 months
* Severe hypoglycemia resulting in seizure or loss of consciousness in the 12 months prior to enrollment
* History of a seizure disorder (except hypoglycemic seizure). Subjects with a history of seizures may be included in the study if they receive written clearance from their neurologist treatment for a seizure disorder
* Coronary artery disease or heart failure. Subjects with a history of coronary artery disease may be included in the study if they receive written clearance from their cardiologist
* Cystic fibrosis
* Active infection
* A known medical condition that in the judgment of the investigator might interfere with the completion of the protocol such as the following examples:

  * Inpatient psychiatric treatment in the past 6 months for either the subject or the subject's primary care giver (i.e., parent or guardian)
  * Presence of a known adrenal disorder
  * Abnormal liver or renal function (Transaminase >2 times the upper limit of normal, Creatinine > 1.5 mg/dL)
  * Active gastroparesis
  * If on antihypertensive, thyroid, anti-depressant or lipid lowering medication, lack of stability on the medication for the past 2 months prior to enrollment in the study
  * Uncontrolled thyroid disease
  * Abuse of alcohol Note: Adequately treated thyroid disease and celiac disease do not exclude subjects from enrollment
* A recent injury to body or limb, muscular disorder, use of any medication, any carcinogenic disease, or other significant medical disorder if that injury, medication or disease in the judgment of the investigator will affect the completion of the exercise protocol
* Current use of a beta blocker medication
* Hematocrit <30% (labs drawn at screening visit or within one month prior to screening for other purposes will suffice for enrollment purposes related to hematocrit)
* Use of pseudoephedrine 48 hours prior to Clinical Research Center (CRC) admission

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2011-03; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Percent of glucose values 71-180 mg/dL of combined day and night readings during the first admission visit | Admission Visit 1
  Group success criterion defined as a mean blood glucose >50%, lower end of one-sided 95% confidence interval >40% and individual criterion of no individual <30%.
Percent of subjects with blood glucose reading of 71-180 mg/dL 4 hours following the breakfast with a missed meal bolus | 4 hours following the breakfast with a missed meal bolus
  Success is defined as >=40% subjects with a blood glucose in the 71-180 mg/dL range.
Percent of subjects with blood glucose reading of 71-180 mg/dL 5 hours following the breakfast with a meal bolus 30% more than the recommended bolus amount | 5 hours following the breakfast with a meal bolus 30% more than the recommended bolus amount
  Success is defined as >=50% subjects with a blood glucose in the 71-180 mg/dL range.
Percent of subjects with a blood glucose nadir <=60 mg/dL following exercise | Following exercise completion
  Success is defined as less than 25% of subjects with a blood glucose nadir <=60 mg/dL.
Overall frequency of hypoglycemia | Includes both admission visits
  Success defined as no subjects with severe hypoglycemia with a low blood glucose resulting in seizure, unconsciousness or the inability to treat oneself.
Overall frequency of hyperglycemia | Includes both admission visits
  Success defined as no subjects with diabetic ketoacidosis (DKA).

SECONDARY OUTCOMES:
Percent of blood glucose values 71-180 mg/dL during the day (9:00AM-11:00PM) of the first admission visit | Admission Visit Day 1 (9:00AM-11:00PM)
  Group success criterion defined as a mean blood glucose >50%, lower end of one-sided 95% confidence interval >40% and individual criterion of no individual <30%.
Percent of blood glucose values 70-180 mg/dL during the night (11:00PM-8:00AM) of the first admission visit | Admission Visit Night 1 (11:00PM-8:00AM)
  Group success criterian defined as a mean blood glucose >60%, lower end of one-sided 95% confidence interval >50% and individual criterion of no individual <30%.
Percent of blood glucose values >400 mg/dL during the first admission visit | Admission Visit 1
  Individual success is defined as no blood glucose values >400 mg/dL.
Percent of blood glucose values <=60 mg/dL during the first admission visit | Admission Visit 1
  No more than 33% of visits with blood glucose <=60 mg/dL
Percent of subjects with a peak blood glucose >400 mg/dL following the breakfast with a missed meal bolus | 4 hours following the breakfast with a missed meal bolus
  Success is defined as less than 5% of subjects have a peak blood glucose >400 mg/dL
Percent of subjects with a nadir blood glucose <=60 mg/dL following the breakfast with a missed meal bolus | 4 hours following the breakfast with a missed meal bolus
  Success is defined as less than 15% of subjects have a nadir blood glucose <=60 mg/dL
Percent of subjects with a peak blood glucose >400 mg/dL following the breakfast with a meal bolus 30% more than the recommended bolus amount | following the breakfast with a meal bolus 30% more than the recommended bolus amount
  Success is defined as less than 5% of subjects have a peak blood glucose >400 mg/dL
Percent of subjects with a nadir blood glucose <=60 mg/dL following the breakfast with a meal bolus 30% more than the recommended bolus amount | following the breakfast with a meal bolus 30% more than the recommended bolus amount
  Success is defined as less than 25% of subjects have a nadir blood glucose <=60 mg/dL

CONTACTS AND LOCATIONS:
Overall Officials: Roy W Beck, MD, PhD, Study Director — Jaeb Center for Health Research; Howard Zisser, MD, Study Chair — Sansum Diabetes Research Institute
Locations (7):
- United States (4):
  - Sansum Diabetes Research Institute, Santa Barbara, California
  - Stanford University, Stanford, California
  - University of Colorado Health Sciences Center- Barbara Davis, Aurora, Colorado
  - University of Virginia, Charlottesville, Virginia
- Montpellier University Hospital, Montpellier, France
- Schneider Children's Medical Center of Israel, Petah Tikva, Israel
- University of Padova, Padua, Italy

REFERENCES:
- [Derived] Chase HP, Doyle FJ 3rd, Zisser H, Renard E, Nimri R, Cobelli C, Buckingham BA, Maahs DM, Anderson S, Magni L, Lum J, Calhoun P, Kollman C, Beck RW; Control to Range Study Group. Multicenter closed-loop/hybrid meal bolus insulin delivery with type 1 diabetes. Diabetes Technol Ther. 2014 Oct;16(10):623-32. doi: 10.1089/dia.2014.0050. Epub 2014 Sep 4. PMID 25188375
- [Derived] Zisser H, Renard E, Kovatchev B, Cobelli C, Avogaro A, Nimri R, Magni L, Buckingham BA, Chase HP, Doyle FJ 3rd, Lum J, Calhoun P, Kollman C, Dassau E, Farret A, Place J, Breton M, Anderson SM, Dalla Man C, Del Favero S, Bruttomesso D, Filippi A, Scotton R, Phillip M, Atlas E, Muller I, Miller S, Toffanin C, Raimondo DM, De Nicolao G, Beck RW; Control to Range Study Group. Multicenter closed-loop insulin delivery study points to challenges for keeping blood glucose in a safe range by a control algorithm in adults and adolescents with type 1 diabetes from various sites. Diabetes Technol Ther. 2014 Oct;16(10):613-22. doi: 10.1089/dia.2014.0066. Epub 2014 Jul 8. PMID 25003311